CLINICAL TRIAL: NCT05252052
Title: Barriers and Facilitators to Long-Acting Reversible Contraception: Perspectives of Adolescents and Healthcare Providers in Rural Haiti
Brief Title: Contraception Perspectives in Adolescents in Haiti
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Abbey Masonbrink, Pediatric Hospitalist, Children's Mercy Hospital Kansas City
Other Study IDs: STUDY00001626
Record Dates: First submitted 2022-01-07; First posted 2022-02-23 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Contraception
MeSH Terms: interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adolescents 14-24 years old: Adolescents 14-24 years old
  Interventions: Other: Interviews/Surveys
- Health care providers in rural Haiti: Health care providers in rural Haiti
  Interventions: Other: Interviews/Surveys

INTERVENTIONS:
Other: Interviews/Surveys — This is a cross sectional survey and interviews of adolescents 14- 18 years old and HCPs living in rural Haiti

SUMMARY:
The overall goal of this study is to assess facilitators and barriers to contraception with a focus on long-acting reversible contraception (LARC) among adolescents and health care providers (HCPs) in rural Haiti. The investigator plans to accomplish the following objectives:

DETAILED DESCRIPTION:
Objective 1: Develop locally-informed surveys and in-depth interview guides, based on the ecologically-expanded Theory of Planned Behavior, to assess attitudes, social norms, perceived behavioral control, and intentions regarding contraception, with a focus on LARC, among adolescents and HCPs in rural Haiti.

Objective 2: Conduct a formative mixed methods study of attitudes, social norms, perceived behavioral control, and intentions regarding contraception, with a focus on LARC, among female adolescents (N=150 survey, 25-50 in-depth interviews) and HCPs (N=15; survey and in-depth interviews) in rural Haiti.

ELIGIBILITY:
Inclusion Criteria:•

* Adolescents who are biologically female and have reproductive potential (14-24 years old)
* Adolescents who reside in the birthing clinic catchment area
* Health care providers, including nurse midwives, who work at the local birthing clinic and providers at the local hospital

Exclusion Criteria:

-Subjects who are determined to have severe psychiatric illness or cognitive impairment (based on research team assessment).

Ages: 14 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Adolescents 14-24 years old and health care providers in rural Haiti
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Identification of facilitators and barriers to contraception use | Data collection will occur over one day for individual participants. Study data collection will occur over 18 months
  The primary outcome is identification of facilitators and barriers to contraception use among adolescent participants based on responses to the eTPB domains described in Table 1. The investigator will also explore facilitators and barriers to contraception use among HCP participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rupe ER, Rodean J, Hurley EA, Miller MK, Boncoeur MD, Masonbrink AR. Menstrual health among adolescents and young adults in rural Haiti. Reprod Health. 2022 Dec 20;19(1):227. doi: 10.1186/s12978-022-01533-4. PMID 36539795
- [Result] Masonbrink AR, Hurley EA, Schuetz N, Rodean J, Rupe E, Lewis K, Boncoeur MD, Miller MK. Sexual behaviors, contraception use and barriers among adolescents and young adults in rural Haiti. BMC Womens Health. 2023 Mar 27;23(1):137. doi: 10.1186/s12905-023-02268-5. PMID 36973773